CLINICAL TRIAL: NCT00459290
Title: A Phase II Evaluation of Mifepristone in the Treatment of Recurrent or Persistent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Mifepristone in Treating Patients With Recurrent or Persistent Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170K
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2014-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mifepristone 200 mg PO daily (Experimental): Mifepristone 200 mg PO daily administered on a continuous basis (every 4 weeks is considered one cycle) until disease progression or adverse effects prohibit further therapy.
  Interventions: Drug: mifepristone

INTERVENTIONS:
Drug: mifepristone

SUMMARY:
RATIONALE: Progesterone can cause the growth of ovarian epithelial cancer , primary peritoneal cancer, or fallopian tube cancer. Hormone therapy using mifepristone may fight ovarian epithelial cancer and primary peritoneal cancer by lowering the amount of progesterone the body makes.

PURPOSE: This phase II trial is studying the side effects and how well mifepristone works in treating patients with recurrent or persistent ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of mifepristone in patients with recurrent or persistent ovarian epithelial, primary peritoneal, or fallopian tube carcinoma.
* Determine the toxicity of this drug in these patients.

Secondary

* Determine the duration of progression-free survival and overall survival of patients treated with this drug.
* Determine the potential impact of platinum sensitivity, initial performance status, and age on prognosis in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral mifepristone once daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube carcinoma*

  * Recurrent or refractory disease NOTE: *Histological confirmation of original primary tumor required
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, and MRI OR ≥ 10 mm by spiral CT scan

  * Must have ≥ 1 target lesion

    * Tumors within a previously irradiated field are designated as nontarget lesions unless progression is documented or a biopsy is obtained to confirm persistence ≥ 90 days after completion of radiotherapy
* Prior treatment with 1 platinum-based chemotherapeutic regimen (comprising carboplatin, cisplatin, or another organoplatinum compound) for management of primary disease required

  * Initial treatment may have included any of the following:

    * High-dose therapy
    * Consolidation therapy
    * Extended therapy administered after surgical or nonsurgical assessment
  * Patients must meet ≥ 1 of the following criteria:

    * Treatment-free interval after platinum therapy of < 12 months
    * Progressed during platinum-based therapy
    * Persistent disease after a platinum-based regimen
* Not eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* No active infection requiring antibiotics
* No other invasive malignancies within the past 5 years, except non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery, radiotherapy, or chemotherapy
* No prior cancer treatment that would preclude protocol therapy
* No prior radiotherapy to any portion of the abdominal cavity or pelvis unless for treatment of ovarian cancer

  * Prior radiotherapy for localized cancer of the breast, head and neck, or skin is permitted, provided it was completed > 3 years prior to study entry and no recurrent or metastatic disease exists
* No prior chemotherapy to any portion of the abdominal cavity or pelvis unless for treatment of ovarian cancer

  * Prior chemotherapy for localized cancer of the breast is permitted, provided it was completed > 3 years prior to study entry and no recurrent or metastatic disease exists
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* At least 2 weeks since other prior hormonal therapy (e.g., testosterone, estrogen, progestin, or gonadotropin-releasing hormone antagonists)
* At least 3 weeks since other prior therapy directed at the malignant tumor, including biological or immunologic agents
* One prior cytotoxic regimen (defined as any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa) for management of recurrent or persistent disease allowed
* No prior non-cytotoxic therapy for management of recurrent or persistent ovarian epithelial or primary peritoneal carcinoma
* No prior mifepristone

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Rocereto, MD, Study Chair — Cancer Institute of New Jersey at Cooper - Voorhees
Locations (22):
- United States (22):
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin

REFERENCES:
- [Result] Rocereto TF, Brady WE, Shahin MS, Hoffman JS, Small L, Rotmensch J, Mannel RS. A phase II evaluation of mifepristone in the treatment of recurrent or persistent epithelial ovarian, fallopian or primary peritoneal cancer: a gynecologic oncology group study. Gynecol Oncol. 2010 Mar;116(3):332-4. doi: 10.1016/j.ygyno.2009.10.071. Epub 2009 Nov 17. PMID 19922989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 5/7/2007 and closed to accrual on 10/29/2007.
Groups:
- Mifepristone: Mifepristone 200 mg PO daily administered on a continuous basis (every 4 weeks considered as one cycle) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Mifepristone
Started | 24
Completed | 19 (Patients treated until disease progression; completed defined as off treatment due to progression.)
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 22
Age, Customized [Number; unit: participants]
  40-49 years | 1
  50-59 years | 6
  60-69 years | 8
  70-79 years | 6
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since study entry, or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
  CT scan or MRI is used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: Every other cycle, for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels.
Population: Eligible and treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 22
percentage of participants | 13.6 [2.9 to 34.9]

2. Primary Outcome: Proportion of Patients With Objective Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Per RECIST v1.0 for target lesions and assessed by MRIor CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  CT scan or MRI is used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: as for outcome 1
Population: Eligible and treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 22
percentage of participants | 4.5 [0.1 to 22.8]

3. Primary Outcome: Number of Participants With Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: Every cycle, during treatment (average of 3 months).
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 22
Participants
  Anemia | 1
  Coagulation | 2
  Dermatologic | 1
  Gastrointestinal | 1
  Hemorrhage | 1

4. Secondary Outcome: Progression-free Survival
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mifepristone
Number analyzed (Participants) | 22
months | 1.8 [1.7 to 3.2]

5. Secondary Outcome: Overall Survival
Time Frame: Five years
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mifepristone
Number analyzed (Participants) | 22
months | NA [7.5 to NA] — NA (not available): insufficient number of participants with events.

6. Secondary Outcome: Progression-free Survival by Platinum Sensitivity
Description: Platinum Senstive defined as treatment free interval >6 months on most recent platinum
Time Frame: as for outcome 1
Population: Eligible and treated participants with treatment free interval available
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Not Platinum Sensitive | Platinum Sensitive
Number analyzed (Participants) | 13 | 8
months | 1.7 [1.7 to 3.8] | 1.9 [1.1 to 4.2]
Statistical Analysis 1: Comparison: Not Platinum Sensitive vs Platinum Sensitive; Test type: Superiority or Other; p = 0.7912, Log Rank

7. Secondary Outcome: Progression-free Survival by Performance Status
Time Frame: as for outcome 1
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- GOG Performance Status 0: Fully active, able to carry on all pre-disease performance without restriction.
- GOG Performance Status 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work.
Arm/Group | GOG Performance Status 0 | GOG Performance Status 1
Number analyzed (Participants) | 13 | 9
months | 1.8 [1.7 to 4.1] | 1.7 [0.9 to 3.2]
Statistical Analysis 1: Comparison: GOG Performance Status 0 vs GOG Performance Status 1; Test type: Superiority or Other; p = 0.1545, Log Rank

8. Secondary Outcome: Progression-free Survival by Age (y)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | < 60 | 60 <70 | >=70
Number analyzed (Participants) | 7 | 8 | 7
months | 1.7 [0.9 to 2.4] | 4.0 [1.6 to 8.1] | 1.7 [1.1 to 1.8]
Statistical Analysis 1: Comparison: < 60 vs 60 <70 vs >=70; Test type: Superiority or Other; p = 0.0648, Log Rank

ADVERSE EVENTS:
Time Frame: every cycle during treatment
Arm/Group | Mifepristone
Serious Adverse Events (participants affected / at risk) | 8/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mifepristone (N=22)
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Perforation, Gi - Colon (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Pain: Abdominal Pain Nos (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mifepristone (N=22)
Neutrophils (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 7
Inr (Vascular disorders) | 2
Fatigue (General disorders) | 9
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hot Flashes (Endocrine disorders) | 4
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Distention (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Anorexia (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 3
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 2
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 3
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 1
Ast (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Bilirubin (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 1
Mood Alteration - Anxiety (Nervous system disorders) | 1
Irritability (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 3
Neuropathy-Motor (Nervous system disorders) | 1
Blurred Vision (Eye disorders) | 2
Pain: Pelvis (General disorders) | 1
Pain: Pleura (General disorders) | 1
Pain: Extremity-Limb (General disorders) | 1
Pain: Back (General disorders) | 1
Pain: Joint (General disorders) | 1
Pain: Bladder (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 7
Pain: Tumor (General disorders) | 1
Pain: Muscle (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Urinary Frequency (Renal and urinary disorders) | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No